CLINICAL TRIAL: NCT05735392
Title: Liquid Biopsy: Intercepting Mutational Trajectories of HER2 Breast Cancer Inpatients Under T-DM1 Treatment
Brief Title: Liquid Biopsy: Intercepting Mutational Trajectories of HER2 (Human Epidermal Growth Factor Receptor 2) Breast Cancer (GIM21 Trial)
Acronym: GIM21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GIM21 - LiqERBcept
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Breast Cancer
Keywords: LiqERBcept; Trastuzumab emtansine; Liquid Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab emtansine as per SmPC for liquid biopsy and tissue collection (Other): Patients will receive trastuzumab emtansine (T-DM1) at 3.6 mg/kg intravenously every 21 days, as perSummary of Product Characteristics (SmPC).
  Peripheral blood samples will be taken by venipuncture prior to initiation of study therapy (T0), and at designated time-points after the first (T1) the second (T2), the third(T3)and after the sixth(T6), the ninth(T9), until the 12thcycle of T-DM1(see Fig.1) on-treatment and finally at progression.
  Interventions: Other: Both blood and tissues collection for patients with metastatic breast cancer HER2+ pretreated with no more than one line of anti-HER2 therapy for advanced breast cancer.

INTERVENTIONS:
Other: Both blood and tissues collection for patients with metastatic breast cancer HER2+ pretreated with no more than one line of anti-HER2 therapy for advanced breast cancer. — Both blood and tissues will be obtained duringT-DM1 treatment of enrolled patients at the participating Sites at the study specific timelines.

SUMMARY:
This is an open, interventional, non-pharmacological, prospective study. Patients will receive trastuzumab emtansine (T-DM1) at 3.6 mg/kg intravenously every 21 days, as per Summary of Product Characteristics (SmPC). This is a no-profit study.

DETAILED DESCRIPTION:
T-DM1 effects will be monitored by a combination of Next Generation Sequencing (NGS, tumor tissue) and Liquid Biopsy (LB, blood), as described below, to capture molecular events (gene aberrations, mainly mutations) associated with (or causative of) relapse as well as primary/adaptive resistance to HER2 blockade.

This study will prospectively monitor these events throughout the clinical history of the patients (archival tissues, blood collection, aimed biopsies). No investigational drugs will be administered.

This protocol is classified as "interventional" for two reasons:

1. dedicated, additional blood drawings (liquid biopsies)are collected in addition to the routine bloodtests being requested as per standard clinical practice;
2. the study involves occasional fine-needle biopsy on accessible (e.g. cutaneous) metastatic foci in selected patients to confirm their HER2 status, as per good medical practice.

These will represent an additional opportunity of targeted NGS.

Both blood (a) and tissues (b) will be obtained during T-DM1 treatment of enrolled patients at the participating Sites at the study specific timelines.

ELIGIBILITY:
Inclusion criteria

1. Male and female patients with a documented diagnosis of metastatic HER2-positive breast cancer (BC) as defined by an immunohistochemistry (IHC) score of 3+, alternatively score 2+ and HER2 amplification ratio ≥ 2.0
2. All patients eligible to treatment with T-DM1, according to SmPC previously treated with a taxane and trastuzumab. Patients who previously underwent first-line treatment with an association of TTZ with PTZ are also eligible. No more than one line of anti-HER2 treatment for advanced disease are allowed.
3. Available tissue from the primary tumor. If possible, newly obtained core or excisional biopsy on metastatic site at baseline (this biopsy won't impact on timing for patient enrollment and not leading to patient exclusion). High quality genomic DNA from the above for NGS mutational analysis.
4. Patients with both measurable and non-measurable disease (according to modified RECIST 1.1 criteria) are eligible.
5. 18 years of age on day of signing informed consent.
6. a left ventricular ejection fraction of 50% or more (determined by echocardiography or multiple-gated acquisition [MUGA] scanning);
7. an Eastern Cooperative Oncology Group performance status of 0 or 1.
8. Adequate organ function (obtained within 14 days prior to treatment study) as evidenced by:

   1. Absolute neutrophil count (ANC) 1.5 X 109/L without myeloid growth factor support for 7 days preceding the lab assessment;
   2. Haemoglobin (Hgb) 9 g/dL (90 g/L); < 9 g/dL (< 90 g/L) is acceptable if hemoglobin is corrected to 9 g/dL (90 g/L) ;
   3. Platelet count 75 X 109/L without blood transfusions for 7 days preceding the lab assessment;
   4. Bilirubin 1.5 X upper limit of normal (ULN), except for patients with a documented history of Gilbert's disease;
   5. Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) 2.5 X ULN (for patients with liver metastases 5 X ULN);
9. Life expectancy > 12 weeks;
10. Written informed consent obtained before any screening procedure and according to local guidelines.

Exclusion criteria

1. Prior treatment with T-DM1.
2. Symptomatic central nervous system (CNS) metastases, or treatment for these metastases within the 2 months preceding enrollment.
3. Current participation in study therapy, or previous participation in a study involving the administration of an investigational agent within 4 weeks of administration of the first dose of treatment.
4. History of symptomatic congestive heart failure or serious cardiac arrhythmia requiring treatment; a history of myocardial infarction or unstable angina within 6 months before.
5. Female patients who are pregnant or lactating, who plan to get pregnant, or who have a positive serum pregnancy test prior to first dose of study treatment.
6. Prior malignancy (other than breast cancer) except for non-melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 5 years prior to enrollment.
7. Any other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation.
8. Patients with psychiatric illness, social situation or geographical situation that would preclude informed consent or limit compliance with study requirements, as determined by the Investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Number of index mutations | About 4 years
  1. Number of index mutations and resistance-associated mutations in the bloodstream. Index mutations are defined as the number of mutation detected in tissue biopsies from either or both the primary lesions and the most recent recurrence, whenever available. Resistance mutations known to arise during non-T-DM1 HER2-blockade include mutations of PIK3CA (phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha), PIK3R1 (Phosphoinositide-3-Kinase Regulatory Subunit 1), AKT1 (AKT1 AKT serine/threonine kinase 1), and EGF1R (Epidermal Growth Factor Receptor 1).These may be a special case of index mutations. Other known genomic aberrations occurring under HER2 blockade and potentially testable in bloodier PTEN (Phosphatase and tensin homolog) loss and overexpression of p95HER2 (p95HER2/611 carboxy terminal fragment), MUC4 (Mucin 4, Cell Surface Associated), and PDK1 (3-Phosphoinositide-dependent kinase 1)
Rate of response/anticipation of relapse | About 4 years
  2. Changes form baseline in thr response rate. First detection of index mutations in blood will be compared with first imaging and medical evidence of relapse (response rate) to determine whether and how the LiqERBcept protocol can lead to earlier detection and improvement in medical care.
Number of de novo mutations | About 4 years
  3. Number of de novo mutations arising during T-DM1 treatment. Few mutations and gene aberrations (see above) are known to associate with primary and acquired resistance to Trastuzumab (TTZ) and Pertuzumab (PTZ), and none is specifically associated with T-DM1 escape, to our knowledge. Possibly, this is due to the rather recent introduction of this antibody-drug conjugate in human therapy.

SECONDARY OUTCOMES:
Number of actionable mutations | About 4 years
  Number of actionable mutations occur during treatment with T-DM1 .

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, MD, Principal Investigator — Clinical issues - Fondazione Policlinico Gemelli; Patrizio Giacomini, Principal Investigator — Central laboratory assesment and liquid biopsy - Oncogenomics and Epigenetics - Istituto Nazionale Tumori "Regina Elena"; Francesco Cognetti, Study Chair — Chairman - Istituto Nazionale Tumori "Regina Elena"
Locations (9):
- Italy (9):
  - A.O. Ospedale Papa Giovanni XXIII - Oncologia, Bergamo
  - I.R.C.C.S. A.O.U San Martino - IST, Genova
  - A.O.U. Policlinico di Modena, Modena
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale S. Cuore Don Calabria, Negrar
  - Fondazione Policlinico Universitario A. Gemelli - Oncologia Medica, Roma
  - Fondazione Policlinico Universitario A. Gemelli - Senologia Oncologica, Roma
  - Istituto Nazionale Tumori "Regina Elena", Roma
  - Policlinico Umberto I, Rome

REFERENCES:
- [Derived] Giordani E, Allegretti M, Sinibaldi A, Michelotti F, Ferretti G, Ricciardi E, Ziccheddu G, Valenti F, Di Martino S, Ercolani C, Giannarelli D, Arpino G, Gori S, Omarini C, Zambelli A, Bria E, Paris I, Buglioni S, Giacomini P, Fabi A. Monitoring changing patterns in HER2 addiction by liquid biopsy in advanced breast cancer patients. J Exp Clin Cancer Res. 2024 Jun 29;43(1):182. doi: 10.1186/s13046-024-03105-9. PMID 38951853